CLINICAL TRIAL: NCT06294743
Title: The Treatment Efficacy of Posterior Tibia Nerve Neuroprolotherapy on Dysmenorrhea
Brief Title: Posterior Tibia Nerve Neuroprolotherapy for Dysmenorrhea
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Jing-Dung, SHEN, Chief Attending, Taichung Armed Forces General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C202304001
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea; Prolotherapy
Keywords: dysmenorrhea; prolotherapy
MeSH Terms: conditions — Dysmenorrhea | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Group-1, posterior tibial nerve neuroprolotherapy will be administered during the first two menstrual cycles, followed by oral acetaminophen (500mg) for the subsequent two menstrual cycles. Conversely.
  Group-2, oral acetaminophen (500mg) will be given during the initial two menstrual cycles, followed by a transition to posterior tibial nerve neuroprolotherapy for the last two menstrual cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Experimental): Posterior tibial nerve neuroprolotherapy will be administered during the first two menstrual cycles, followed by oral acetaminophen (500mg) for the subsequent two menstrual cycles
  Interventions: Procedure: Posterior tibial nerve neuroprolotherapy; Drug: Acetaminophen 500Mg Tab
- Group-2 (Experimental): Oral acetaminophen (500mg) will be given during the initial two menstrual cycles, followed by a transition to posterior tibial nerve neuroprolotherapy for the last two menstrual cycles.
  Interventions: Procedure: Posterior tibial nerve neuroprolotherapy; Drug: Acetaminophen 500Mg Tab

INTERVENTIONS:
Procedure: Posterior tibial nerve neuroprolotherapy — Real-time ultrasound guided needle injecting 10ml of 5% dextrose solution around the posterior tibial nerve to elicit a neurostimulatory response.
Drug: Acetaminophen 500Mg Tab — Oral acetaminophen 500mg tab stat, followed by Q6h if needed.

SUMMARY:
The goal of this crossover study is to assessed the treatment efficacy of posterior tibia nerve neuroprolotherapy on dysmenorrhea. The primary outcome is the improvement of Visual Analogue Scale. The main question it aims to answer is:

•Could the posterior tibial nerve neuroprolotherapy alleviate the pain of dysmenorrhea.

Participants will be randomly allocated into two groups, Group-1 will receive neuroprolotherapy in the first 2 menstrual cycles followed by oral acetaminophen(500mg) for the subsequent 2 menstrual cycles. Group02 will received oral acetaminophen(500mg) in initial 2 menstrual cycles, followed by receiving neuroprolotherapy for the subsequent 2 menstrual cycles.

DETAILED DESCRIPTION:
This trial is a crossover study involving the enrollment of 60 women aged 20-50 who experience normal menstrual cycles accompanied by menstrual pain. These participants will be randomly allocated into two distinct groups. In Group-1, posterior tibial nerve neuroprolotherapy will be administered during the first two menstrual cycles, followed by oral acetaminophen (500mg) for the subsequent two menstrual cycles. Conversely, in Group-2, oral acetaminophen (500mg) will be given during the initial two menstrual cycles, followed by a transition to posterior tibial nerve neuroprolotherapy for the last two menstrual cycles. The primary outcome measure for this trial is the improvement in the Visual Analog Scale (VAS). Secondary outcomes include an assessment of changes in quality of life before and after treatment, as evaluated using the SF-36 questionnaire. Furthermore, pulse diagnosis instruments will be employed to analyze alterations in meridian energy before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50 who experience normal menstrual cycles accompanied by menstrual pain

Exclusion Criteria:

* Malignant tumors requiring treatment.
* Pregnant
* Those who have other acute and chronic pain and are receiving relevant drug treatment.
* Those who are allergic to acetaminophen or have contraindications.
* Those who use hormonal contraceptives at the same time.
* Those with coagulation disorders or taking anticoagulant drugs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The patients who suffered with dysmenorrhea.
Enrollment: 60 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline, 1st month,2nd month,3rd month,4th month.
  The visual analogue scale ranged from 0(no pain) to 10(severe pain)

SECONDARY OUTCOMES:
The SF-36v2® Health Survey | Baseline, 1st month,2nd month,3rd month,4th month.
  The SF-36 questionnaire is a short-form health survey that measures each of the following eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each health domain score contributes to the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Armed Forces General Hospital, Taichung, Other (Non US), Taiwan

IPD SHARING:
Plan to Share IPD: No